CLINICAL TRIAL: NCT02630680
Title: A Multicentre, European, Observational, Drug Utilisation Study (DUS) of BLI800 (Eziclen®/Izinova®) as a Bowel Cleansing Preparation
Brief Title: Eziclen Drug Utilisation in Real Life Setting
Acronym: DUS-BLI800
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: 8-79-58800-001; EUPAS9361 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Bowel Cleansing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colorectal diseases patients
  Interventions: Drug: Eziclen®/Izinova®

INTERVENTIONS:
Drug: Eziclen®/Izinova®

SUMMARY:
The purpose of the study is to assess Eziclen/Izinova drug utilisation in the real life setting in a representative sample of the European target population.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for a prescription of BLI800 (Eziclen®/Izinova®) as a cleansing bowel preparation in accordance with the marketing authorisation.
* Patient having provided written informed consent.

Exclusion Criteria:

* Patient not eligible for a prescription of BLI800 (Eziclen®/Izinova®) as a cleansing bowel preparation in accordance with the marketing authorisation. Specifically, patients in whom there is a contraindication for use of this product, including patients with congestive heart failure, severe renal insufficiency of active inflammatory bowel disease, are not eligible for inclusion in this study.
* Patient being prescribed a cleansing bowel preparation other than BLI800 (Eziclen®/Izinova®).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal diseases patients from specialised gastroenterology, hepatogastroenterology departments ("referral centres") and endoscopy departments ("non referral centres").
Sampling Method: Probability Sample
Enrollment: 1286 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
Volume of liquid intake | on the day of the colonoscopy
  Assessment of non-compliance in terms of insufficient liquid intake. The volume of water and clear liquids taken will be derived from the remaining volumes as recorded on the patient's leaflet and reported by the Investigator. Compliance to the hydration guidelines expressed in terms of a ratio (actual volume taken versus theoretical volume).

SECONDARY OUTCOMES:
Number of adverse events | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (16):
- Czechia (3):
  - Ustredni vojenska nemocnice, Prague
  - Krajská zdravotní, a.s., nemocnice Teplice, Teplice
  - Ústeckoorlická nemocnice, Ústí nad Orlicí
- Germany (8):
  - MVZ Ortenau Achern, Innere Medizin, Achern
  - Gemeinschaftspraxis Dres. Klausmann, Aschaffenburg
  - Klinikum Aschaffenburg-Alzenau, Standort Aschaffenburg, Aschaffenburg
  - Chefarzt der Medizinischen Klinik III, Westpfalz Klinikum GmbH, Standort I Kaiserslautern, Kaiserslautern
  - MVZ Innere Medizin Marburg, Dres. Drude und Partner, Marburg
  - Medizinisches Versorgungszentrum, Münster
  - Praxisgemeinschaft Innere am Stadtpark, Nuremberg
  - Gastro-Praxis Wiesbaden (Gastrodata), Wiesbaden
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - Elisabeth-Tweesteden Ziekenhuis, Tilburg
- Poland (3):
  - Copernicus Medical Entity, Gdansk
  - Instytut Medycyny, Lublin
  - Oncology center - Institutte, Warsaw